CLINICAL TRIAL: NCT03912012
Title: Endothelial Dysfunction Could be an Early Biomarker of Renal Impairment in Children and Adolescent With Type 1 Diabetes. Pilot Study DiaDEP
Brief Title: Pilot Study DiaDEP
Acronym: DiaDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0518
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1; Type1diabetes
Keywords: Diabetes mellitus type 1; Type 1 diabetes; diabetes; pediatrics; Glomerular hyperfiltration; endothelial dysfunction; children; adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children and adolescent with a history of type 1 diabetes (Other): Children and adolescent from 10 to 18 years old, with a history of type 1 diabetes for at least 10 years. Glomerular hyper filtration and endothelial dysfunction will be evaluate.
  Interventions: Drug: Iohexol renal clearance measurement; Device: microcirculation assessment through Laser Doppler associated to iontophoresis.; Device: Cardiovascular assessment though Intima-media Thickness and Extra-media Thickness measurement; Biological: Blood sampling; Biological: Urine sampling; Device: High-resolution peripheral quantitative computed tomography (HR-pQCT); Radiation: Dual-energy X-ray (DXA)

INTERVENTIONS:
Drug: Iohexol renal clearance measurement — intravenous injection of Iohexol (Omnipaque 300mg) with blood sampling at 0, 120, 180 and 240 minutes (during Day 1.
Device: microcirculation assessment through Laser Doppler associated to iontophoresis. — endothelial function evaluated following a protocol of iontophoresis of acetylcholine (during Day 1).
Device: Cardiovascular assessment though Intima-media Thickness and Extra-media Thickness measurement — carotid ultrasound (during Day 1)
Biological: Blood sampling — 37 mL of blood sample will be performed at Day 1
Biological: Urine sampling — The urinary collection will be done during the Day 1, on the first morning urination
Device: High-resolution peripheral quantitative computed tomography (HR-pQCT) — assessment of the Body Mass Index by HR-pQCT (during the Day 1)
Radiation: Dual-energy X-ray (DXA) — assessment of bone parameters by DXA (during the Day 1)

SUMMARY:
With an increased incidence of pediatric type 1 diabetes (T1D) and a decrease in age at diagnosis, children are exposed to complications such as renal impairment at a very young age.

The current biomarker used to diagnose renal impairment is microalbuminuria, but it's a late marker. Early screening is a major issue to reduce T1D consequences.

Early glomerular hyperfiltration (GHF) could participate in the development and progression of nephropathy. Hyperfiltration has also been associated with a systemic endothelial dysfunction and with changes in arterial stiffness, suggesting, at least to a certain extent, a state of generalized vascular dysfunction.

Diabetes is responsible for very early neurovascular dysfunctions, detectable with techniques to evaluate cutaneous neurovascular interaction. Those should help bringing to light very early microcirculation impairment, particularly precocious endothelial dysfunction (ED).

No study about correlation between GHF and ED is currently available. The hypothesis assessed is those of a strong correlation between ED and GHF in children and adolescent with a story of T1D for at least 10 years.

This pilot study should allow assessing ED's and GHF's proportions in our population, in order to conduct a larger study to prove, in a prospective way, the prognostic value of ED in the apparition of nephropathy, taking into count other factors such as diabetes duration or stability.

This measure could be included in the global evaluation of microangiopathy risk in children and then take action to prevent negative outcomes.

The second aspect of this study is the assessment of other functions and metabolisms possibly impaired in T1D: osseous microarchitecture, vitamin D status and precocious evaluation of macro angiopathy through intima media thickness measurement.

Long term diabetes in children is associated with shorter and leaner bones, despite a correct mineralization, a reduced bone density and a fracture risk increased six fold. Bone status in the population will be evaluated through the study of bones microarchitecture via HR-pQCT (High Resolution peripheral Quantitative Computed Tomography) on both tibia and radius, dual-energy X-ray absorptiometry (DXA), and bone turn over biochemical markers.

Results on bone microarchitecture in a preexisting cohort of healthy children and adolescents will be used to compare results.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 10 et < 18 years old
* Type 1 diabetes diagnosed more than 10 years previously.
* Written informed consent signed by both parents or legal representatives, child or adolescent's agreement.
* Health cover

Exclusion Criteria:

* Associated pathology with a potential impact on cutaneous microcirculation or renal function.
* Aspirin or other non-steroid anti-inflammatory treatment with potential impact on endothelial function in the 3 weeks preceding the visit.
* Examination with injection of contrast agent during the last 48 hours
* Smoking
* Ongoing pregnancy or breast feeding
* Hypersensitivity to acetylcholine
* Contraindication to Iohexol
* Ongoing treatment with growth hormone, non-inhaled corticosteroids or anti-calcineurins;
* History of treatment with oral corticosteroids (not inhaled) more than 3 successive months regardless of seniority;
* Paracetamol treatment less than a week old;

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Glomerular hyper filtration (Glomerular filtration > 135 mL/min/1,73 m2) | Day 1
  assessed through Iohexol renal clearance measurement

SECONDARY OUTCOMES:
Endothelial function in the forearm. | Day 1
  Endothelial function will be evaluated by the microcirculation assessment through Laser Doppler associated to iontophoresis of acetylcholine.
Intima media thickness | Day 1
  The intima media thickness will be performed by Echo Doppler of both right and left common carotid
arterial blood pressure | Day 1
  arterial blood pressure measurement
Bone mass | Day 1
  Bone mass will be performed by Dual-energy X-ray absorptiometry (DXA) on both spine and whole body.
bone density | Day 1
  bone density will be performed by Dual-energy X-ray absorptiometry (DXA) on both spine and whole body.
quantization of bone mineral content | Day 1
  quantization of bone mineral content will be performed by Dual-energy X-ray absorptiometry (DXA) on both spine and whole body.
Volumetric compartmental density | Day 1
  Volumetric compartmental density will be performed by High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) on radius and tibia (Right tibia and non-dominant arm radius). (Unless there is a history of fracture for one of those bones, in which case the opposite side will be studied instead.)
trabecular microarchitecture | Day 1
  trabecular microarchitecture will be performed by High Resolution peripheral Quantitative Computed Tomography (HR-pQCT) on radius and tibia (Right tibia and non-dominant arm radius). (Unless there is a history of fracture for one of those bones, in which case the opposite side will be studied instead.)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant - Groupement Hospitalier Est, Bron, France